CLINICAL TRIAL: NCT04875819
Title: Safety and Immunogenicity Following Meningococcal and Pneumococcal Immunization Among Adult People Living With HIV: A Single Center, Non-blinded, Randomized Clinical Trial
Brief Title: Safety and Immunogenicity Following Meningococcal and Pneumococcal Immunization Among Adult People Living With HIV
Acronym: MENPI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, Clinical professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-19001166; 2020-000863-22 (EudraCT Number)
Record Dates: First submitted 2021-04-12; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Hiv; Meningococcal Infections; Pneumococcal Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningococcal Infections; Pneumococcal Infections | interventions — Meningococcal Vaccines; 4CMenB vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menveo + Bexsero (Experimental)
  Interventions: Drug: Neisseria meningitidis oligosaccharide conjugate vaccine and recombinant protein-based vaccine
- Prevenar13 + Pneumovax23 (Experimental)
  Interventions: Drug: 13 valent pneumococcal conjugate vaccine and 23 valent pneumococcal polysaccharide vaccine

INTERVENTIONS:
Drug: Neisseria meningitidis oligosaccharide conjugate vaccine and recombinant protein-based vaccine — One dose (0.5 ml) of conjugate vaccine against meningococcal serogroups ACWY (Menveo®) and one dose of a recombinant protein-based vaccine against meningococcal serogroup B (Bexsero®) at day 0 followed by another dose (0.5 ml) of each vaccine at day 60.
  Other Names: Menveo® and Bexsero®
  Arms: Menveo + Bexsero
Drug: 13 valent pneumococcal conjugate vaccine and 23 valent pneumococcal polysaccharide vaccine — One dose (0.5 ml) of pneumococcal conjugate vaccine (Prevenar13®) at day 0 and one dose (0.5 ml) of pneumococcal polysaccharide vaccine (Pneumovax23®) at day 60.
  Other Names: Prevenar13® and Pneumovax23®
  Arms: Prevenar13 + Pneumovax23

SUMMARY:
MENPI is an investigator-initiated single-centre randomized controlled trial which aims to assess the efficacy and safety of meningococcal and pneumococcal vaccination in adults living with HIV receiving antiretroviral treatment.

Participants are randomized 1:1 to either a two-dose Menveo® and Bexsero® regimen or a Prevenar13®/Pneumovax23® prime-boost regimen at day 0 and day 60 and cross over on day 90. All participants will follow an identical follow up program including plasma collection, pharyngeal swab, and adverse event registration.

Immunogenicity will be determined on venous blood sampled at 30 days post-vaccination and yearly for five years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Seropositive for HIV-1
* Recipient of ART
* Plasma HIV-RNA < 500 copies/ml
* Patients written consent obtained

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of meningococcal or pneumococcal vaccination
* Allergies towards any of the vaccine components
* Temperature > 38 ᵒC
* Sign of bacterial infection
* Previous known or suspected disease caused by N. meningitidis
* Active AIDS associated illness
* Active malignancy
* End-stage renal or liver disease
* Bleeding disorder
* Recipient of any blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within the last month
* Use of immunosuppressive agents (corticosteroids, cancer chemotherapeutic agents etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in immunogenic response from baseline, Menveo | Day 30 and year 1, 2, 3, 4, and 5 post-vaccination
  A ≥4-fold rise in rabbit complement source (rSBA) for the four serogroups A, C, Y, and W-135. Seroprotection is defined as an rSBA titre ≥1:8 and patients will be classified as previously immune if baseline rSBA is ≥1:8.
Change in immunogenic response from baseline, Bexsero | Day 30 and year 1, 2, 3, 4, and 5 post-vaccination
  A ≥4-fold rise in antibody titers against a panel of four meningococcal serogroup B reference strains between pre-vaccination and post-vaccination timepoints, or a post-vaccination antibody titre ratio of ≥1:4 for individuals who were seronegative before vaccination.
Change in immunogenic response from baseline, Prevenar13/Pneumovax23 | Day 30 and year 1, 2, 3, 4, and 5 post-vaccination
  A ≥2-fold rise in serum anti-capsular IgG GMC for 12 shared pneumococcal polysaccharides (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F)

SECONDARY OUTCOMES:
Number of participants with immediate adverse events | 30 minutes post-vaccination
Number of participants with short term adverse events | Day 5 post vaccination
Number of participants with long term adverse events | Day 90 post-vaccination
Streptococcus pneumoniae carriage rates | Baseline and day 30 post-vaccination
  Proportion of study subject with a culture or PCR positive pharyngeal swab sample
Neisseria meningitidis carriage rates | Baseline and day 30 post-vaccination
  Proportion of study subject with a culture or PCR positive pharyngeal swab sample

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Tinggaard, M.D., Principal Investigator — Department of Infectious Diseases, Hvidovre Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Background] Miller L, Arakaki L, Ramautar A, Bodach S, Braunstein SL, Kennedy J, Steiner-Sichel L, Ngai S, Shepard C, Weiss D. Elevated risk for invasive meningococcal disease among persons with HIV. Ann Intern Med. 2014 Jan 7;160(1):30-7. doi: 10.7326/0003-4819-160-1-201401070-00731. PMID 24166695
- [Background] Simmons RD, Kirwan P, Beebeejaun K, Riordan A, Borrow R, Ramsay ME, Delpech V, Lattimore S, Ladhani S. Risk of invasive meningococcal disease in children and adults with HIV in England: a population-based cohort study. BMC Med. 2015 Dec 9;13:297. doi: 10.1186/s12916-015-0538-6. PMID 26654248
- [Background] Harboe ZB, Larsen MV, Ladelund S, Kronborg G, Konradsen HB, Gerstoft J, Larsen CS, Pedersen C, Pedersen G, Obel N, Benfield T. Incidence and risk factors for invasive pneumococcal disease in HIV-infected and non-HIV-infected individuals before and after the introduction of combination antiretroviral therapy: persistent high risk among HIV-infected injecting drug users. Clin Infect Dis. 2014 Oct 15;59(8):1168-76. doi: 10.1093/cid/ciu558. Epub 2014 Jul 17. PMID 25038114
- [Background] MacNeil JR, Rubin LG, Patton M, Ortega-Sanchez IR, Martin SW. Recommendations for Use of Meningococcal Conjugate Vaccines in HIV-Infected Persons - Advisory Committee on Immunization Practices, 2016. MMWR Morb Mortal Wkly Rep. 2016 Nov 4;65(43):1189-1194. doi: 10.15585/mmwr.mm6543a3. PMID 27811836
- [Background] Lujan-Zilbermann J, Warshaw MG, Williams PL, Spector SA, Decker MD, Abzug MJ, Heckman B, Manzella A, Kabat B, Jean-Philippe P, Nachman S, Siberry GK; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1065 Protocol Team. Immunogenicity and safety of 1 vs 2 doses of quadrivalent meningococcal conjugate vaccine in youth infected with human immunodeficiency virus. J Pediatr. 2012 Oct;161(4):676-81.e2. doi: 10.1016/j.jpeds.2012.04.005. Epub 2012 May 22. PMID 22622049
- [Background] Frota ACC, Ferreira B, Harrison LH, Pereira GS, Pereira-Manfro W, Machado ES, de Oliveira RH, Abreu TF, Milagres LG, Hofer CB. Safety and immune response after two-dose meningococcal C conjugate immunization in HIV-infected children and adolescents in Rio de Janeiro, Brazil. Vaccine. 2017 Dec 15;35(50):7042-7048. doi: 10.1016/j.vaccine.2017.10.043. Epub 2017 Oct 31. PMID 29100708
- [Background] Pedersen RH, Lohse N, Ostergaard L, Sogaard OS. The effectiveness of pneumococcal polysaccharide vaccination in HIV-infected adults: a systematic review. HIV Med. 2011 Jul;12(6):323-33. doi: 10.1111/j.1468-1293.2010.00892.x. Epub 2010 Nov 8. PMID 21059168
- [Background] Lee KY, Tsai MS, Kuo KC, Tsai JC, Sun HY, Cheng AC, Chang SY, Lee CH, Hung CC. Pneumococcal vaccination among HIV-infected adult patients in the era of combination antiretroviral therapy. Hum Vaccin Immunother. 2014;10(12):3700-10. doi: 10.4161/hv.32247. PMID 25483681
- [Background] Sogaard OS, Schonheyder HC, Bukh AR, Harboe ZB, Rasmussen TA, Ostergaard L, Lohse N. Pneumococcal conjugate vaccination in persons with HIV: the effect of highly active antiretroviral therapy. AIDS. 2010 Jun 1;24(9):1315-22. doi: 10.1097/QAD.0b013e328339fe0b. PMID 20559037
- [Background] Rodriguez-Barradas MC, Serpa JA, Munjal I, Mendoza D, Rueda AM, Mushtaq M, Pirofski LA. Quantitative and Qualitative Antibody Responses to Immunization With the Pneumococcal Polysaccharide Vaccine in HIV-Infected Patients After Initiation of Antiretroviral Treatment: Results From a Randomized Clinical Trial. J Infect Dis. 2015 Jun 1;211(11):1703-11. doi: 10.1093/infdis/jiu819. Epub 2014 Dec 23. PMID 25538270